CLINICAL TRIAL: NCT01660841
Title: A Multicenter, Open-label, Phase III Study to Determine the Safety and Efficacy of Gadobutrol 1.0 Molar in Japanese Subjects Referred for Contrast-enhanced MRI of the Central Nervous System (CNS)
Brief Title: Safety and Efficacy of Gadobutrol 1.0 Molar in Japanese Subjects for CNS Imaging
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16260
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Magnetic Resonance Imaging
Keywords: Magnetic resonance imaging; central nervous system; contrast media; gadobutrol
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Gadobutrol (Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadovist, BAY86-4875) — A single bolus injection of gadobutrol 1.0M 0.1mmol/kg body weight.

SUMMARY:
Purpose of the study is to look at the safety (what are the side effects) and efficacy (how well does it work) of gadobutrol when used for taking images of the brain and spine. The results of the Magnetic Resonance Imaging (MRI) will be compared to the results of images taken without contrast (gadobutrol).

ELIGIBILITY:
Inclusion Criteria:

* Subjects referred for a contrast-enhanced Magnetic Resonance Imaging (MRI) of the central nervous system based on current clinical symptoms or results of a previous imaging procedure

Exclusion Criteria:

* Subjects with any contraindication to the MRI examination
* Subjects with severe renal disease to end stage renal disease
* Subjects scheduled or are likely to require a biopsy or any interventional therapeutic procedure within 72 (±4) hours after the study MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Scores for visualization parameter: degree of contrast enhancement | Day of gadobutrol injection (Day 0)
  Blinded readers evaluate contrast of at maximum 5 lesions and 4 normal brain structures in scans taken with and without injection of gadobutrol on a 4-point-scale.
Scores for visualization parameter: border delineation | Day of gadobutrol injection (Day 0)
  Blinded readers evaluate border delineation of at maximum 5 lesions and 4 normal brain structures in scans taken with and without injection of gadobutrol on a 4-point-scale.
Scores for visualization parameter: internal morphology | Day of gadobutrol injection (Day 0)
  Blinded readers evaluate internal morphology of at maximum 5 lesions and 4 normal structures in scans taken with and without gadobutrol on a 3-point-scale.
Number of detected lesions | Day of gadobutrol injection (Day 0)
  Blinded readers determine number of detected lesions in scans with and without gadobutrol.

SECONDARY OUTCOMES:
Percentage of exact match of the MRI diagnosis with the final clinical diagnosis | Day of gadobutrol injection (Day 0)
  An exact match is defined as identical diagnosis given by the blinded reader and the independent standard of truth committee.
Sensitivity and specificity to detect abnormal/normal brain tissue | Day of gadobutrol injection (Day 0)
  Blinded readers classify the brain tissue as normal or abnormal based on the MRI sets.
Sensitivity and specificity to detect malignant Central Nervous System(CNS) lesions | Day of gadobutrol injection (Day 0)
  Percentage to correctly detect presence and absence of malignant lesions which are derived from the MR diagnosis of readers when compared with the diagnosis of the independent standard of truth committee.
Number of participants with treatment emergent adverse events as a measure of safety and tolerability | 3 days after injection (Day 3)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Japan (13):
  - Nagoya, Aichi-ken
  - Funabashi, Chiba
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Fukuyama, Hiroshima
  - Kobe, Hyōgo
  - Fujisawa, Kanagawa
  - Kawasaki, Kanagawa
  - Yokohama, Kanagawa
  - Daitō, Osaka
  - Kishiwada, Osaka
  - Shimonoseki, Yamaguchi
  - Ube, Yamaguchi